CLINICAL TRIAL: NCT01948453
Title: Effect of Garlic Tablet on Carotid Intima Media Thickness and Flow-mediated Dilation in Patients Undergoing Angioplasty
Brief Title: Effect of Garlic Tablet Some Indicators Related to Atherosclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Dr., Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 513
Record Dates: First submitted 2013-09-14; First posted 2013-09-23 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2013-09

CONDITIONS: Coronary Artery Disease
Keywords: CAD; CIMT; FMD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Garlic (Active Comparator): daily consumption of two odor controlled garlic tablets
  Interventions: Dietary Supplement: Garlic
- Placebo (Placebo Comparator): daily consumption of placebo

INTERVENTIONS:
Dietary Supplement: Garlic — Garlic tablet in adjunct to medical treatment
  Arms: Garlic

SUMMARY:
The purpose of this study is to determine whether garlic in adjunct to conventional medical treatment is effective in improving carotid intima media thickness (CIMT), Flow mediated dilation (FMD) and plasma lipid profile or c-reactive protein of coronary artery disease (CAD) patients.

ELIGIBILITY:
Inclusion Criteria:

* angiography confirmed coronary artery disease
* lack of consistent use of the garlic in the last month

Exclusion Criteria:

Change in type of medication during study

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Carotid Intima Media Thickness | 12 weeks
  Change from baseline and compared to placebo group in Carotid Intima Media Thickness at 12 weeks

SECONDARY OUTCOMES:
Flow-mediated dilatation | 12 weeks
  Change from baseline and compared to placebo group in Flow-mediated dilatation at 12 weeks

OTHER OUTCOMES:
plasma levels of Alanine Aminotransferase, Aspartate Aminotransferase, creatinine, lipid profile, C-Reactive Protein | 12 weeks
  Change from baseline in plasma levels at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Javad Nasrollahzadeh, Ph.D., Study Chair — Department of Clinical Nutrition and Diet Therapy, National Nutrition and Food Technology Research Institute, Faculty of Nutrition Sciences and Food Technology, Shahid Beheshti University of Medical Sciences; Ali Z Mehr, M.D., Study Director — Department of Cardiology, Rajaei Cardiovascular, Medical & Research Center; Marjan M Roshan, Ph.D., Principal Investigator — Department of Clinical Nutrition and Diet Therapy, National Nutrition and Food Technology Research Institute, Faculty of Nutrition Sciences and Food Technology, Shahid Beheshti University of Medical Sciences
Locations (1):
- Rajaei Cardiovascular, Medical & Research Center, Tehran, Iran